CLINICAL TRIAL: NCT00488098
Title: An Open Label, Randomized, Parallel Groups, Bioequivalence Study to Compare a Single Oral Dose of GSK372475B or GSK372475C in Male and Female Healthy Volunteers.
Brief Title: GSK372475 Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SND110117
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Depressive Disorder
Keywords: Healthy Bioequivalence
MeSH Terms: conditions — Depressive Disorder | interventions — GSK372475

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK372475

SUMMARY:
The study is to show the new salt formulation of GSK372475 is equivalent to the old salt formulation of GSK372475.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males/Females aged 18-45 years
* Non-smokers
* BMI 19-30 kg.m2
* QTc<450msec

Exclusion Criteria:

* Use of oral contraception
* Positive breath alcohol and drug screen
* Regular alcohol consumption
* Current psychiatric illness or within 1 year.
* History of GI, hepatic or renal disease
* Uncontrolled hypertension

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2007-07

PRIMARY OUTCOMES:
GSK372475 plasma level at AUC0-72, AUC0-inf, CMax and TMax | at predose, 0.5,1-24, 36,48,60,72,96 and 1-4 weeks post dose.

SECONDARY OUTCOMES:
Adverse events | all visits
vitals (all visits) + ECG | at screening,Day-1, predose, 1,6,24,48,72 and week 2 post dose.
labs | at screening and 2 weeks post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Toronto, Ontario, Canada